CLINICAL TRIAL: NCT05511233
Title: OutComes of Implementing EnhAnced Recovery AftEr Intestinal Surgery Protocol in Newborns: CARES Study
Brief Title: ERAS Protocol in Newborns: CARES Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Katip Celebi University (Other)
Responsible Party: Principal Investigator, ESRA ARDAHAN AKGUL, Assistant Professor, Principal Investigator, Izmir Katip Celebi University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 2022
Record Dates: First submitted 2022-08-02; First posted 2022-08-22 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-10

CONDITIONS: Pediatric
Keywords: pediatric surgery; enhanced recovery
MeSH Terms: interventions — Postoperative Period

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CONTROL GROUP (No Intervention): Control Group: Electronic health records of the newborns who do not receive breast milk in the first 48 hours of the postoperative period will be in the control group.
- ERAS GROUP (Experimental): ERAS Group: Electronic health records of the newborns who had breastmilk within the first 48 hours in the postoperative period will be in the ERAS group.
  Interventions: Dietary Supplement: feeding with breastmilk within 48 hours after surgery

INTERVENTIONS:
Dietary Supplement: feeding with breastmilk within 48 hours after surgery — Electronic health records of babies who feed and not fed with breastmilk within 48 hours after surgery
  Arms: ERAS GROUP

SUMMARY:
Aim: To determine whether the enteral feeding time and the type of the nutrient (according to the ERAS Recommendations) have any effect on LoS, complications, body weight gain, time until oral feeding, and time until first stool who have undergone intestinal surgery.

Design: A blinded, retrospective, randomized controlled trial. Setting: One-centred. Participants: Newborns who had intestinal surgery in the Ege University Faculty of Medicine Hospital Neonatal Surgery Intensive Care Unit and whose records can be accessed retrospectively from the electronic health records will be included. Those whose early enteral feeding initiation is contraindicated will not be included in the study.

DETAILED DESCRIPTION:
Every year, approximately 1.7 million children, most of them in low- and middle-income countries, are deprived of safe and evidence-based surgical and anaesthesia practices in the world, resulting in lifelong disability or mortality. The care of children who have undergone surgery, and especially newborns, has different physiological and sociological difficulties compared to adults. Newborns make up a particularly complex patient population due to their blood volume, temperature imbalance, immature immune systems, nutritional needs for growth and recovery, and inability to communicate. Therefore, guidelines have been developed to improve perioperative care and recovery through research, education, supervision and implementation of evidence-based practices in newborns. One of these guidelines is Perioperative Care in Neonatal Intestinal Surgery by Enhanced Recovery After Surgery® (ERAS) Society. In this guideline, there are recommendations on surgical practices, antimicrobial prophylaxis, hypothermia, perioperative fluid management, perioperative analgesia, optimal haemoglobin level, perioperative communication, postoperative nutritional care, mucous fistula refeeding and parental involvement. Among these recommendations, the initiation of early feeding (in the first 48 hours) is one of the core elements of nursing care. In patients who are not contraindicated such as necrotizing enterocolitis and volvulus, early feeding has effects on length of hospital stay (LoS), risk of wound infection, and increasing C-reactive protein levels. Although studies support this recommendation, different clinical conditions may require a delay in feeding, therefore, evidence for this recommendation was found to be weak in the guideline. Studies in different populations are needed to increase the strength of this recommendation. Also, the nutrient content is as important as the time of initiation of feeding, because thanks to its anti-infectious effect, it reduces the incidence of respiratory and gastrointestinal tract infections and necrotizing enterocolitis. Some studies have also shown neurodevelopmental advantages and a reduced incidence of metabolic disease. In addition, it has been determined that breast milk provides proper growth in newborns who have undergone surgery and prevents postoperative complications in babies who have had heart surgery. Therefore, in the ERAS protocol, it is recommended that the first preferred nutrient is breast milk. In the postoperative period, feeding intolerances can be seen in newborns as a complication because due to the operation, a dilated proximal segment may occur with hypoplasia of the smooth muscle or enteric nervous system, which leads to feeding intolerance. To prevent this complication, it is considered appropriate to use breast milk, which is a nutrient with high tolerability and can support intestinal adaptation thanks to its barrier function, probiotics and immunoglobulins it contains.

Design: A blinded, retrospective, randomized controlled trial. Setting: One-centred. Participants: Newborns who had intestinal surgery in the Ege University Faculty of Medicine Hospital Neonatal Surgery Intensive Care Unit and whose records can be accessed retrospectively from the electronic health records will be included. Those whose early enteral feeding initiation is contraindicated will not be included in the study.

Groups:

ERAS Group: Newborns who had breastmilk within the first 48 hours in the postoperative period will be in the ERAS group.

Control Group: Newborns who do not receive breast milk in the first 48 hours of the postoperative period will be in the control group.

Variables: The dependent variables of this study are the length of hospital stay, time until full feed (120 ml/kg/day), time until first oral feeding, time until first stool, body weight gain, feeding intolerance (abdominal distention and repeated vomiting-more than three times a day) and Accordion Severity Grading System of Surgical Complications Score. The independent variables of this research are the type of the surgery, enteral feeding time and the type of the nutrient.

Randomization: It was found that 80 newborns met the inclusion criteria for the control group. To randomly select 21 of these 80 newborns Random Integer Generator on www.random.org will be used. (https://www.random.org/integers/?num=21&min=1&max=80&col=1&base=10&format=html&rnd=new) It was found that 65 newborns met the inclusion criteria for the ERAS group. To randomly select 21 of these 65 newborns Random Integer Generator on www.random.org will be used (https://www.random.org/integers/?num=21&min=1&max=65&col=1&base=10&format=html&rnd=new). No stratification will be used in randomization.

Main Outcomes and Measures: The main outcomes of this study are LoS, time until full feed (120 ml/kg/day), time until first oral feeding, time until first stool, body weight gain, feeding intolerance (abdominal distention and vomiting). The secondary outcome is the Accordion Severity Grading System of Surgical Complications Score20.

Accordion Severity Grading System of Surgical Complications Score: It was developed by Strasberg in 2009. In this scoring, the frequency of complications is evaluated under the sub-headings of mild complications, moderate complications, severe complications requiring intervention with or without anaesthesia, organ system failure or death.

Statistics: The minimum sample size in each group was considered 21 and a total of 42 using a power formula with a = 0.05, power of 95%, and 0.50 effect size 1.06. To calculate the sample size G*Power 3.1.9.2 programme was used. In determining the differences between the groups in terms of the main outcomes, the Mann-Whitney U or Chi-square tests will be used since they are independent groups.

ELIGIBILITY:
Inclusion Criteria:

* Newborns who had intestinal surgery in the Ege University Faculty of Medicine Hospital Neonatal Surgery Intensive Care Unit and
* whose records can be accessed retrospectively from the electronic health records will be included.

Exclusion Criteria:

* Those whose early enteral feeding initiation is contraindicated will not be included in the study.

Ages: 1 Day to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 42 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Length of Stay | 14 days
  Time from surgery to discharge
full feed | through study completion, an average of 14 days
  time until full feed (120 ml/kg/day)
first oral feeding | through study completion, an average of 14 days
  time until first oral feeding
first stool | through study completion, an average of 14 days
  time until first stool
body weight gain | through study completion, an average of 14 days
  body weight gain
feeding intolerance | through study completion, an average of 14 days
  abdominal distention and repeated vomiting-more than three times a day

SECONDARY OUTCOMES:
the Accordion Severity Grading System of Surgical Complications Score | 14 days
  It was developed in 2009. In this scoring, the frequency of complications is evaluated under the sub-headings of mild complications, moderate complications, severe complications requiring intervention with or without anaesthesia, organ system failure or death

CONTACTS AND LOCATIONS:
Overall Officials: Esra ARDAHAN AKGÜL, Asst. Prof., Study Chair — İzmir Katip Çelebi University

IPD SHARING:
Plan to Share IPD: No